CLINICAL TRIAL: NCT04683835
Title: Evaluation of Cognitive State in Senior Subjects Using Neurosteer Single-channel EEG With an Interactive Assessment Tool
Brief Title: Evaluation of Cognitive State in Senior Subjects Using Neurosteer EEG System
Status: Completed | Type: Observational
Sponsor: Neurosteer Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 092020
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognition; Neurology; EEG; Neurosteer
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients: Patients who are assessed by the clinical staff using Mini-Mental State Exam (MMSE)
  Interventions: Device: Neurosteer Aurora system

INTERVENTIONS:
Device: Neurosteer Aurora system — The system is composed of hardware and software modules that facilitate the capture and interpretation of electrophysiological data as well as enable viewing the processed data in real time and offline. An electrode patch is attached on the subject's forehead to capture the electrophysiological signal. The signal is sent via low energy Bluetooth to an EEG Monitor. The signal is then sent via Wi-Fi to the cloud where the data is stored on a HIPAA compliant server. Data analysis performed in the cloud transforms the electrophysiological signal into easily readable data of brain activity, which is accessible via any web interface

SUMMARY:
This is an observational study. Patients who fulfill all inclusion criteria and none of the exclusion criteria will be enrolled in the study, be neurologically evaluated and will go through EEG recordings while listening to an auditory cognitive assessment tool. EEG recordings will be analyzed using proprietary computational analyses.

DETAILED DESCRIPTION:
One of the major problems in the prevention and treatment of neurological disorders, is the lack of cost effective and reliable tools to assess neurodegeneration on a large scale at a very early stage. Although current imaging methods give a clear image of the brain atrophy involved in neurodegenerative disorders, there are deficiencies prohibiting their usage for prevention-scanning of large high-risk population such as high price, long set-up time and the need for trained personnel to conduct the test. Therefore, the development of a reliable tool to assess brain neurodegeneration, associated with cognitive decline independent of personal interpretation and/or variance between clinicians and between medical facilities would be highly valuable. This tool would allow the healthcare team to make appropriate treatment decisions that could aid in neurodegenerative disease prevention.

The Neurosteer system provides objective neurological biomarkers using a wearable easy-to-use affordable system. The system facilitate the capture and interpretation of EEG data with only a single patch of electrodes, attached on the subject's forehead. Neurosteer examination includes completing auditory tasks while measuring brain activity with the device. The data is analyzed using machine learning methods to produce biomarkers, enabling a report of the patient's activity in real time and offline. The examination is easy to preform and can be conducted in every clinic or in patients' homes.

In this study, clinical staff will identify potential subjects and will examine the eligibility of subject according to inclusion and exclusion criteria. Research staff will inform the patient on study's objective and design. Patients will sign the Informed Consent Form (ICF). Research staff will set up an initial session using the Neurosteer system. In this session the patient will perform auditory cognitive assessment tasks. The patient will be re-examined in the same experimental setting over the next 7 days and at least 1 day later. Level of cognition will be assessed by the Neurosteer technology.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 50.
* MMSE ≥ 24.
* Patient is able to collaborate.
* No other cognitive comorbidity.
* No seizure events.

Exclusion Criteria:

* MMSE < 24.
* Any verbal or non-verbal form of objection from patient or form patient's family member or significant other.
* Presence of several cognitive comorbidity.
* Damage to integrity of scalp and/or skull.
* Skin irritation in the facial and forehead area.
* Significant hearing impairments.
* History of drug abuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients from the inpatient rehabilitation department at Dorot Geriatric Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ady Sasson, Dr., Principal Investigator — Dorot, Geriatric Medical Center
Locations (1):
- Dorot - Netanya Geriatric Medical Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Guerrero-Berroa E, Luo X, Schmeidler J, Rapp MA, Dahlman K, Grossman HT, Haroutunian V, Beeri MS. The MMSE orientation for time domain is a strong predictor of subsequent cognitive decline in the elderly. Int J Geriatr Psychiatry. 2009 Dec;24(12):1429-37. doi: 10.1002/gps.2282. PMID 19382130
- [Background] Meir-Hasson Y, Kinreich S, Podlipsky I, Hendler T, Intrator N. An EEG Finger-Print of fMRI deep regional activation. Neuroimage. 2014 Nov 15;102 Pt 1:128-41. doi: 10.1016/j.neuroimage.2013.11.004. Epub 2013 Nov 15. PMID 24246494
- [Background] Meir-Hasson Y, Keynan JN, Kinreich S, Jackont G, Cohen A, Podlipsky-Klovatch I, Hendler T, Intrator N. One-Class FMRI-Inspired EEG Model for Self-Regulation Training. PLoS One. 2016 May 10;11(5):e0154968. doi: 10.1371/journal.pone.0154968. eCollection 2016. PMID 27163677
- [Background] Goldway N, Ablin J, Lubin O, Zamir Y, Keynan JN, Or-Borichev A, Cavazza M, Charles F, Intrator N, Brill S, Ben-Simon E, Sharon H, Hendler T. Volitional limbic neuromodulation exerts a beneficial clinical effect on Fibromyalgia. Neuroimage. 2019 Feb 1;186:758-770. doi: 10.1016/j.neuroimage.2018.11.001. Epub 2018 Nov 5. PMID 30408596
- [Background] Keynan JN, Cohen A, Jackont G, Green N, Goldway N, Davidov A, Meir-Hasson Y, Raz G, Intrator N, Fruchter E, Ginat K, Laska E, Cavazza M, Hendler T. Electrical fingerprint of the amygdala guides neurofeedback training for stress resilience. Nat Hum Behav. 2019 Jan;3(1):63-73. doi: 10.1038/s41562-018-0484-3. Epub 2018 Dec 10. PMID 30932053

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.86 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 80
MMSE score [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) is a structured assessment tool that evaluates cognitive functioning.
  The MMSE produces a total possible score ranging from 0 to 30. Patients who score below 24 would typically be suspected for cognitive decline or early dementia.
  units on a scale | 27.21 (2.05)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Cognition Level Changes as Evaluated by Current Clinical Tools (i.e. MMSE) and Brain Activity Features Extracted Using the Neurosteer Technology.
Description: Cognition level changes will be evaluated by:
  1. Mini Mental State Examination (MMSE). A commonly used assessment tool that evaluates cognitive functioning and produces a total possible score of 30 points. Patients who score below 24 are typically suspected of cognitive decline.
  2. Neurosteer system (single channel EEG recording during cognitive auditory tasks). Using data analysis (a variant of the wavelet packet analysis and the best basis algorithm), the EEG signal is transformed into brain activity features (e.g. ST4, A0).
  Pearson correlation will be calculated between the mean activity of the EEG features and individual's MMSE score.
Time Frame: MMSE score will be taken from previous evaluation performed in the institute. Through study completion, brain activity features will be assessed twice within 7 days using the Neurosteer EEG system.
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Patients
Number analyzed (Participants) | 80
Pearson correlation coefficient | 0.1486

2. Secondary Outcome: Inter-patient Variability Between Two Consecutive Measurement Sessions.
Description: One limitation in the pilot study was high variability among subjects. Therefore, the aim of this study is to evaluate within-patient variability. For this purpose, subjects in this study will undergo two consecutive assessments over a period of one week.
  The within-patient variability will be evaluated by calculating the Pearson correlation between the mean activity of the EEG features in the first assessment session and the mean activity of the EEG features in the second assessment session.
Time Frame: Through study completion, the brain activity features of each subject will be assessed twice within 7 days, using the Neurosteer EEG system.
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Patients
Number analyzed (Participants) | 80
Pearson correlation coefficient | 0.583

ADVERSE EVENTS:
Time Frame: Through study completion, twice a week during EEG recordings, up to 1 year.
Description: In this study the risk for any Serious Adverse Events is low, as the nature of the experiment is entirely non-invasive and merely records EEG data.
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04683835/Prot_SAP_000.pdf